CLINICAL TRIAL: NCT06332417
Title: Combined Effects of Ba-Duan-Jin Based Deep Breathing Exercises and Forced Expiratory Technique in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Combined Effects of Ba-Duan-Jin Based Deep Breathing Exercises and Forced Expiratory Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0364
Record Dates: First submitted 2024-03-04; First posted 2024-03-27 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary disease; Breathing Exercises; Ba-Duan Jin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Ba-Duan-Jin Exercise + FET (Forced Expiratory Technique)
  Interventions: Other: Ba-Duan-Jin Based Deep Breathing Exercises
- Control Group (Active Comparator): FET (Forced Expiratory Technique) only
  Interventions: Other: FET (Forced Expiratory Technique)

INTERVENTIONS:
Other: Ba-Duan-Jin Based Deep Breathing Exercises — Pressing Up to the Heavens: Deep inhales while raising arms, promoting lung expansion.
  Drawing the Bow to Shoot the Eagle: Stretching exercises to improve flexibility and posture.
  Arms: Intervention group
Other: FET (Forced Expiratory Technique) — The forced expiratory technique sometimes referred to as a 'huff', is used to help force secretions (phlegm) up the throat so it can be removed via the mouth without the pain of coughing.
  Arms: Control Group

SUMMARY:
This study will be a randomized control trial. A total of 68 patients will be recruited and randomly assign to the experimental group or the control group in a 1:1 ratio. Participants in the experimental group will receive a 8-week Ba-duan jin exercise training intervention along with Forced Expiratory Technique at least 3 days a week and 30 minutes a day, while participants in the control group will be only given Forced Expiratory intervention and will be told to maintain their original lifestyle for 8 weeks along with standard COPD treatment.

DETAILED DESCRIPTION:
This study will be a randomized control trial. A total of 68 patients will be recruited and randomly assign to the experimental group or the control group in a 1:1 ratio. Participants must have a documented diagnosis of Chronic Obstructive Pulmonary Disease (COPD) based on established clinical criteria (such as GOLD guidelines). Participants should be between 40 and 55 years old. Participants should be in a stable condition, free from exacerbations or respiratory infections for at least four weeks prior to the study enrollment. Participants in the experimental group will receive a 8-week Ba-duan jin exercise training intervention along with Forced Expiratory Technique at least 3 days a week and 30 minutes a day, while participants in the control group will be only given Forced Expiratory intervention and will be told to maintain their original lifestyle for 8 weeks along with standard COPD treatment. All participants will continue with their prescribed medication. During this study time participants will be given instructions on how to perform the prescribed pulmonary exercises. After each exercise session the FEV1 and exercise capacity of the patients will be checked.

ELIGIBILITY:
Inclusion Criteria:

* Both Genders
* Diagnosis of COPD: Participants must have a documented diagnosis of Chronic Obstructive Pulmonary Disease (COPD) based on established clinical criteria (such as GOLD guidelines)
* Participants should be between 40 and 55 years old
* Participants should be in a stable condition, free from exacerbations or respiratory infections for at least four weeks prior to the study enrollment.
* Participants must be physically able to participate in Ba-Duan-Jin based deep breathing exercises.

Exclusion Criteria:

* Individuals with significant comorbidities such as asthma, pulmonary fibrosis, bronchiectasis, or lung cancer
* Participants with severe cardiovascular conditions, such as recent myocardial infarction, unstable angina, or uncontrolled hypertension, which could limit exercise participation
* Individuals with severe cognitive impairment or psychiatric conditions preventing them from understanding and following the exercise program
* Individuals with severe physical impairments unrelated to COPD, hindering their ability to perform exercises or assessments.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
36-Item Short Form Survey (SF-36) | 8 Weeks
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study for the objective measure of the quality of life.
  It comprises 36 questions that cover eight domains of health:
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to high QOL
FEV1/FVC ratio | 8 Weeks
  The FEV1/FVC ratio is the ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs. The normal value for this ratio is above 0.75-85, though this is age dependent.
Exercise Tolerance : 6 minute walk test | 8 Weeks
  a patient can quickly walk back and forth in a 30-m (100-foot) corridor in a period of 6 min, referred to as the 6-min walk distance (6MWD).
Forced vital capacity (FVC) | 8 Weeks
  Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible. It's measured by spirometry , which is a common breathing test to check lung function.
Forced expiratory volume (FEV1) | 8 Weeks
  Forced expiratory volume (FEV1) calculates the amount of air that a person can force out of their lungs in 1 second. It's measured by spirometry , which is a common breathing test to check lung function.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Faizan Hamid, MS-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Social Security Teaching Hospital, Lahore, Punhab, Pakistan

IPD SHARING:
Plan to Share IPD: No